CLINICAL TRIAL: NCT04908774
Title: Effects of Repetitive Cycles of a Fasting Mimicking Diet on Sperm Quality in Men Between 18 and 60 With Reduced Sperm Quality According to the WHO-5 Criteria.
Brief Title: Effects of a Fasting Mimicking Diet on Sperm Quality
Acronym: KiWu-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KiWu-B
Record Dates: First submitted 2021-05-10; First posted 2021-06-01 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Sub Fertility, Male; Fertility Disorders; Sperm Count, Low
Keywords: fasting; natural therapies; fasting mimicking diet; caloric restriction; dietary restriction; dietary intervention; lifestyle modification; spermiogram; sperm motility; liquefaction time; sperm morphology; total sperm count; sperm density
MeSH Terms: conditions — Infertility, Male; Oligospermia; Fasting | interventions — Angptl4 protein, mouse; Diet Therapy

STUDY DESIGN:
Intervention Model Description: This explorative study is conducted in form of a randomized, controlled trial design with a fasting intervention and a waiting list, which continues the usual diet.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to mask a fasting intervention for the participant or the study personel. Therefore only outcome assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting Mimicking Diet Group (Experimental): The intervention group follows a fasting mimicking diet for 5 days every 6-8 weeks (a total of 3 times in 5 months).
  Interventions: Behavioral: Fasting Mimicking Diet
- Control Group (No Intervention): This group maintains their individual diet during the whole time of the study. After 6 months they are offered a fasting intervention.

INTERVENTIONS:
Behavioral: Fasting Mimicking Diet — The mobile application "Salufast" provides standardised fasting packages for 5 days of approx. 500 kcal and accompanies the participants during all fasting days.
  Other Names: Fasting; Dietary Intervention
  Arms: Fasting Mimicking Diet Group

SUMMARY:
This study investigates the effect of repetitive cycles of a Fasting Mimicking Diet (3x5 days in six months) on sperm quality in men

DETAILED DESCRIPTION:
This 2-arm, randomized, controlled exploratory clinical trial aims to explore fasting as a novel supportive treatment in male infertility due to reduced sperm quality according to WHO5-criteria. The participants will be randomized in two groups. The intervention group follows a regime of a periodic fasting mimicking diet (3x5 days in six months, every 6-8 weeks, accompanied via a mobile application), whereas the patients on the waiting list continue their normal diet. Spermiograms are taken about every 2 months following the WHO-5 criteria. In addition, qualitative interviews will be conducted including individual and focus group interviews with a subgroup of participants.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 60 years
* Unfulfilled desire to have a child > 1 year
* reduced sperm quality (proven via spermiogram according tho WHO-5 criteria)
* informed consent
* 20 kg/m² <= BMI <= 35 kg/m²

Exclusion Criteria:

* No sufficient communication possible
* severely impairing cognitive illness
* serious mental illness
* Patients with anatomical/organic damage of reproductive organs
* Eating disorders in the medical history
* Serious internal diseases
* Lack of internet access
* No consent to randomisation
* Participation in other studies

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — biological male sex
Enrollment: 22 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Total sperm motility | change from baseline to 6 months after baseline
  WHO-5 spermiogram parameter to measure sperm quality
Qualitative interview analysis | up to 48 weeks after fasting intervention
  individual and focus group interviews

SECONDARY OUTCOMES:
spermiogram following the WHO-5 criteria | baseline and approx. every 2 months over the course of a year (12 months)
  WHO-5 measurement of sperm quality
quality of life according to the WHO-Five Well-Being Index | baseline, after one week, after 8 (±2) weeks, after 12 (±2) weeks, after 17 (±2) weeks, after 26 (±2) weeks and after 52 (±2) weeks
  WHO-5 questionnaire, validated questionnaire to evaluate the quality of life. It includes 5 questions that assess feelings or moods over the past two weeks. The items in this questionnaire are scaled on a six-point scale. The 5 items result in a total score from a minimum of zero to a maximum of 25, whereby a total score of less than 13 or a score of zero as an answer to one of the questions indicates a possible depression.
mindfulness | baseline, after one week, after 8 (±2) weeks, after 12 (±2) weeks, after 17 (±2) weeks, after 26 (±2) weeks and after 52 (±2) weeks
  MAAS-questionnaire, validated questionnaire to examine mindfulness. It consists of 14 items with four-point Likert scales (never, almost never, sometimes, often, very often). A sum score is formed by adding them up.
anxiety and depression | baseline, after one week, after 8 (±2) weeks, after 12 (±2) weeks, after 17 (±2) weeks, after 26 (±2) weeks and after 52 (±2) weeks
  HADS-questionnaire, validated questionnaire to examine anxiety and depression. The HADS-D is used to assess anxiety and depression in patients with physical diseases or (possibly psychogenic) physical complaints. It measures the degree of anxiety and depressive symptoms during the past week by means of self-report, which is recorded on two subscales with seven items each. The total score can be used as a measure of general psychological impairment.
current mood | baseline, after one week, after 8 (±2) weeks, after 12 (±2) weeks, after 17 (±2) weeks, after 26 (±2) weeks and after 52 (±2) weeks
  ASTS-questionnaire, validated questionnaire to examine current mood.The "Profile of Mood States" served as the basis for the contruction. The ASTS comprises 19 items on five subscales: sadness, hopelessness, fatigue, anger and positive mood.
experienced stress | baseline, after one week, after 8 (±2) weeks, after 12 (±2) weeks, after 17 (±2) weeks, after 26 (±2) weeks and after 52 (±2) weeks
  Cohen-stress scale, validated questionnaire to examine experienced stress. Cohen Perceived Stress Scale (CPSS): The CPSS measures the degree of acute subjective experience of stress (Cohen 1983). It consists of 14 items with four-point Likert scales (never, almost never, sometimes, often, very often). A sum score is formed by summing up the items.
physical fitness | baseline, after one week, after 8 (±2) weeks, after 12 (±2) weeks, after 17 (±2) weeks, after 26 (±2) weeks and after 52 (±2) weeks
  questionnaire to examine physical fitness
Changes in diet | baseline, after one week, after 8 (±2) weeks, after 12 (±2) weeks, after 17 (±2) weeks, after 26 (±2) weeks and after 52 (±2) weeks
  questionnaire to examine diet
quality of relationship | baseline, after one week, after 8 (±2) weeks, after 12 (±2) weeks, after 17 (±2) weeks, after 26 (±2) weeks and after 52 (±2) weeks
  questionnaire to examine the relationship between the two partners desiring to have a child
psychological stress caused by the unfulfilled desire to have children | baseline, after one week, after 8 (±2) weeks, after 12 (±2) weeks, after 17 (±2) weeks, after 26 (±2) weeks and after 52 (±2) weeks
  questionnaire to examine the psychological stress caused by the unfulfilled desire to have children
gratitude | baseline, after one week, after 8 (±2) weeks, after 12 (±2) weeks, after 17 (±2) weeks, after 26 (±2) weeks and after 52 (±2) weeks
  validated questionnaire to examine gratitude
self-efficacy | baseline, after one week, after 8 (±2) weeks, after 12 (±2) weeks, after 17 (±2) weeks, after 26 (±2) weeks and after 52 (±2) weeks
  ASKU, validated questionnaire to examine self-efficacy. The ASKU with three items is used for the economic measurement of subjective competence expectations. It includes the psychological variables self-esteem, internal locus of control, global life satisfaction, optimism as well as the personality traits neuroticism and extraversion from the five-factor model

OTHER OUTCOMES:
liver sonography | up to 14 days before, during and up to 14 days after a fasting intervention
  sonography in a subgroup
reported pregnancy of female partner | up to 12 months after baseline
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Hochschulambulanz für Naturheilkunde der Charité-Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: after the end of the study for 5 years
Access Criteria: on demand